CLINICAL TRIAL: NCT02617979
Title: Improving Mental and Physical Health and Decreasing Hospital Readmission After Pancreatectomy Through Enhanced Patient and Caregiver Education and Engagement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients are receiving detailed packet from department and do not feel they need to go online for additional support.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201511067
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: SAFECARE at Home (Experimental): * Patients randomized to the intervention arm will be assigned a username and password to access a SAFECARE at Home account via the internet. They will also be emailed a link to the site with their username and password.
  * The investigators have worked directly with SAFECARE at Home to create customized lessons for patients undergoing pancreatectomy. These lessons are comprehensive and encompass preoperative preparation as well as postoperative recovery and care. This includes videos, printed material, web-based material, and modules that focus on the pre-treatment, treatment, and follow-up care of patients undergoing surgery for pancreatic cancer.
  * All patients will receive standard pre- and post-operative instructions and care. This will include verbal education about the procedure by the surgeon as well as standard educational patient handouts, which are routinely provided preoperatively to pancreatectomy patients.
  Interventions: Other: SAFECARE at Home customized lessons
- Arm 2: Standard of Care (No Intervention): -All patients will receive standard pre- and post-operative instructions and care. This will include verbal education about the procedure by the surgeon as well as standard educational patient handouts, which are routinely provided preoperatively to pancreatectomy patients.

INTERVENTIONS:
Other: SAFECARE at Home customized lessons
  Arms: Arm 1: SAFECARE at Home

SUMMARY:
The study of readmission is in its infancy in the surgical world, and there are no prospective studies, to the investigators' knowledge, evaluating the efficacy of interventions on preventing readmission following pancreatectomy. Undoubtedly, patients and their caregivers will play a key role in any useful intervention to reduce readmission. Therefore, the investigators' approach is to target perioperative education and engagement of patients and their caregivers in the postoperative recovery of pancreatectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for major pancreatectomy (i.e., pancreaticoduodenectomy, total pancreatectomy, or a distal pancreatectomy).
* At least 18 years of age.
* Able to read and understand English (the SAFECARE at Home program is only implemented in English)
* Has internet access.
* Knowledge of the internet and how to use web-based programs.
* Not pregnant or breastfeeding.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of the SAFECARE at Home program as measured by readmission rate | 30 days
  -The investigators hypothesize that the SAFECARE at HOME program intervention will reduce readmission by half (i.e. from 22% to 11%). The investigators will include a total of 225 evaluable patients in the study, randomized in a 2:1 ratio (i.e. 2 patients in the SAFECARE arm for every 1 patient in the standard of care arm). The designed sample size will allow 80% at a 1-sided alpha=0.1 to detect a 50% decrease in 30-day readmission.

SECONDARY OUTCOMES:
Effect of the SAFECARE at Home program as measured by the number of follow-up visits | Through 30 day post-discharge
  -Follow-up visits include emergency room visits, urgent care visits, unscheduled surgeon office visits, and office calls.
Comparison of quality of life between SAFECARE at Home patients and patients who received standard post-operative care and education as measured by SF-36 | Up to 6 months post-discharge
  -The quality of life as measured by SF-36 (overall and sub-scales) will be summarized using descriptive statistics for each arm and compared by two-way ANOVA for repeated measurement data.
  The Short Form (36) Health Survey (SF-36) is a 36-item, patient-reported survey of patient health.
  -The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan C Fields, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu